CLINICAL TRIAL: NCT01226849
Title: An Open-Label, Pilot Study To Investigate Feasibility and Safety Of Using Bortezomib, Rituximab, Ifosfamide, Carboplatin, Etoposide As Salvage Regime In Previously Treated Patients With Diffuse Large B-Cell Lymphoma
Brief Title: Feasibility Study Of Adding Bortezomib to R-ICE Chemotherapy To Treat Relapsed/ Refractory Diffuse Large B-Cell Lymphoma
Acronym: SGH652
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGH652
Record Dates: First submitted 2010-10-19; First posted 2010-10-22 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2017-04

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: diffuse large B-cell lymphoma relapse refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Bortezomib; Rituximab; Etoposide; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): bortezomib, rituximab, ifosphamide, etoposide, carboplatin
  Rituximab 375mg/m2 day 1 Etoposide 100mg/m2 day 1-3 Carboplatin AUC (5) max 800 days 2 Ifosfamide continuous infusion + Mesna 5/m2/24hr day2 Bortezomib 1.3mg/m2 days 1,4,8,11 G-CSF (SC) recommended
  Interventions: Drug: bortezomib, rituximab, ifosphamide, etoposide, carboplatin

INTERVENTIONS:
Drug: bortezomib, rituximab, ifosphamide, etoposide, carboplatin — Rituximab 375mg/m2 day 1 Etoposide 100mg/m2 day 1-3 Carboplatin AUC (5) max 800 days 2 Ifosfamide continuous infusion + Mesna 5/m2/24hr day2 Bortezomib 1.3mg/m2 days 1,4,8,11 G-CSF (SC) recommended
  Other Names: velcade,; rituxan,; mabtera

SUMMARY:
Incorporation of rituximab to conventional chemotherapy (R-CHOP) has revolutionalized the frontline treatment of diffuse large B-cell lymphoma (DLBCL), one of the commonest subtype of lymphoma. Although the majority of patients are cured, there still remains a substantial number patients (20-30%) who will relapse despite upfront R-CHOP therapy. Recent studies have informed that in the rituximab era, the ability to salvage patients with relapsed DLBCL with the conventional salvage regimens like R-ICE or R-DHAP is significantly poorer than expected. For a patients who has been exposed to rituximab in the frontline, the response rate of conventional salvage chemotherapy is now a mere 51% (Coral Study). This suggests that relapses after rituximab exposure are more severe, strongly implying the presence of rituximab-resistant disease in additional to the selection of more aggressive subtypes of DLBCL which R-CHOP may not have a significant impact on. As R-CHOP is currently the frontline standard of care, more has to be done to augment the current available salvage regimens as a response rate of 51% is unacceptable.

Incorporation of agents targeting rituximab-resistance and also the more aggressive subtype of DLBCL ( ABC subtype) is prudent in the salvage regimen. Bortezomib, a targeted novel agent has potent anti-tumor effects on its own. It has also been show clinically to be able to overcome the adverse risk conferred by the ABC subtype of DLBCL. In addition, preclinical studies have also demonstrated that bortezomib may enhance the biologic activity of rituximab through upregulation of CD20, the target of rituximab.

The investigators hypothesize that adding bortezomib to salvage regimen of DLBCL will be more efficacious. Increasing the response rate will then allow more eligible patients to go on to autologous stem cell transplantation. The investigators intend to test the tolerability and efficacy of the combination of bortezomib with the R-ICE regimen, and attempt to correlate responses with histopathological and gene expression studies of tumor specimens.

DETAILED DESCRIPTION:
The most commonly used regimen for relapsed/refractory diffuse large B-cell lymphoma (DLBCL) is the R-ICE regime (rituximab, ifosphamide, cisplatin and etoposide). It was previously reported to give an overall response rate (RR) of close to 70%, and a complete response rate of 53%. As most DLBCL patients are now treated in the frontline with R-CHOP regimen, the validity of RRs with R-ICE needs to be reevaluated. Results of the CORAL study, a prospective randomized phase III trial comparing R-DHAP vs R-ICE in relapsed DLBCL were recently presented. It was shown that there was no difference in RR between R-ICE and R-DHAP. However, the RR of patients who had received prior rituximab in the frontline setting was significantly lower at 51%, compared with rituximab-naïve patients at 83%. This suggests that relapses after rituximab exposure are more severe. In addition to the risk of more aggressive subtype of DLBCL (activated B-cell [ABC]) that may not be abrogated by rituximab, the presence of rituximab-resistant disease is also strongly implicated. As R-CHOP is currently the frontline standard of care, more has to be done to augment the current available salvage regimens. Incorporation of agents targeting the activated B-cell (ABC)subtype and rituximab-resistance is prudent in the salvage regimen. Bortezomib, a proteosome inhibitor impacts on many cellular processes relevant to the pathogenesis of DLBCL, including inhibition of nuclear factor-kappa B. Preclinical studies have also demonstrated that bortezomib displayed significant antitumor activity against various lymphomas, and in particular the ABC subtype of DLBCL. It is also capable of enhancing the biologic activity of rituximab through upregulation of CD20 in preclinical studies. Demonstration of synergism in these 2 agents, in part due to their dependence on overlapping pathways, suggests that they should be explored as a combination.

On this basis, the investigators aim to conduct a pilot study of adding intravenous bortezomib to R-ICE as a salvage regime for adult patients with relapsed/refractory DLBCL.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven diffuse large B-cell lymphoma in first relapse after CR, less than PR or PR to first line treatment De Novo DLBCL, DLBCL arising from transformed follicular lymphoma or chronic lymphocytic leukaemia are allowed.

   Prior rituximab is allowed Prior radiation is allowed Prior autologous stem cell transplant is allowed CD20 negative relapses are allowed
2. Age between 21-70
3. Written informed consent
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
5. Minimum life expectancy of 3 months
6. Previously treated with chemotherapy containing anthracyclines and rituximab
7. Negative urine or serum pregnancy test on females of childbearing potential
8. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study.
9. Male subject agrees to use an acceptable method for contraception for the duration of the study.
10. No CNS involvement
11. Measurable disease on CT scan by international working group response criteria

Exclusion Criteria:

1. Prior allogeneic transplantation
2. Prior treatment with bortezomib
3. Concomitant use of any other anti-cancer therapy
4. Concomitant use of any other investigational agent
5. Known infection with human immunodeficiency virus (HIV)
6. Patient has known clinically active hepatitis B (carriers of hepatitis B are permitted to enter the study)
7. Contraindication to any drug contained in chemotherapy regimens
8. Not previously treated with anthracycline-containing regimens
9. Impaired liver, renal or other organ function not caused by lymphoma, which will interfere with the treatment schedule
10. Poor bone marrow reserve (neutrophils <1.0 x 109/L or platelets <75 x 10(9)/L unless related to bone marrow infiltration
11. Subject has a calculated or measured creatinine clearance of <20 mL/minute within 14 days before enrollment.
12. Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at Screening has to be documented by the investigator as not medically relevant.
13. Clinically significant active infection
14. Subject has ≥grade 2 peripheral neuropathy or grade 1 with pain within 14 days before enrollment.
15. Patients who are pregnant or breast-feeding
16. Coexistent second malignancy or history of prior malignancy within previous 3 years (excluding non-melanoma skin tumors or in situ carcinoma of the cervix)
17. Any significant medical or psychiatric condition that might prevent the patient from complying with all study procedures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
To evaluate number of participants with adverse events with R-ICE plus bortezomib (VR-ICE) | 2 years
  To evaluate the feasibility, safety and maximum tolerated dose (MTD) of R-ICE plus bortezomib (VR-ICE) in previously treated patients with DLBCL.

SECONDARY OUTCOMES:
Response rate | 2 years
  Response rate at the end of 3 cycles of induction chemotherapy treatment will be assessed. The ability of stem cells mobilization with the regimen and the engraftment rate will also be studied. Lastly, Time to progression or relapse and overall survival will be determined. Biomarkers assessment & correlation of response to subtype DLBCL will be attempted.

CONTACTS AND LOCATIONS:
Overall Officials: Yeow Tee Goh, MBBS MMed, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Gisselbrecht C, Glass B, Mounier N, Singh Gill D, Linch DC, Trneny M, Bosly A, Ketterer N, Shpilberg O, Hagberg H, Ma D, Briere J, Moskowitz CH, Schmitz N. Salvage regimens with autologous transplantation for relapsed large B-cell lymphoma in the rituximab era. J Clin Oncol. 2010 Sep 20;28(27):4184-90. doi: 10.1200/JCO.2010.28.1618. Epub 2010 Jul 26. PMID 20660832
- [Background] Czuczman MS, Olejniczak S, Gowda A, Kotowski A, Binder A, Kaur H, Knight J, Starostik P, Deans J, Hernandez-Ilizaliturri FJ. Acquirement of rituximab resistance in lymphoma cell lines is associated with both global CD20 gene and protein down-regulation regulated at the pretranscriptional and posttranscriptional levels. Clin Cancer Res. 2008 Mar 1;14(5):1561-70. doi: 10.1158/1078-0432.CCR-07-1254. PMID 18316581
- [Background] Dunleavy K, Pittaluga S, Czuczman MS, Dave SS, Wright G, Grant N, Shovlin M, Jaffe ES, Janik JE, Staudt LM, Wilson WH. Differential efficacy of bortezomib plus chemotherapy within molecular subtypes of diffuse large B-cell lymphoma. Blood. 2009 Jun 11;113(24):6069-76. doi: 10.1182/blood-2009-01-199679. Epub 2009 Apr 20. PMID 19380866